CLINICAL TRIAL: NCT00552188
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of the Effect of VIA-2291, a 5-Lipoxygenase Inhibitor, on Vascular Inflammation in Patients After an Acute Coronary Syndrome Event
Brief Title: Phase 2 Study in Vascular Inflammation on Patients After an Acute Coronary Syndrome Event
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tallikut Pharmaceuticals, Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other); Icahn School of Medicine at Mount Sinai (Other); University of Massachusetts, Worcester (Other); Winthrop University Hospital (Other); Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIA-2291-03
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Atherosclerosis
MeSH Terms: conditions — Acute Coronary Syndrome; Atherosclerosis | interventions — atreleuton

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VIA-2291 (Experimental): VIA-2291 100mg
  Interventions: Drug: VIA-2291
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIA-2291 — 100 mg, oral dosing, 1 time daily for 24 weeks
  Arms: VIA-2291
Drug: Placebo — oral dosing, 1 time daily for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of VIA-2291 as compared to placebo on vascular inflammation following 24 weeks of dosing.

DETAILED DESCRIPTION:
The effect of VIA-2291 on vascular inflammation will be assessed through 18FDG PET vascular imaging measurements and various biomarkers after 24 weeks.

ELIGIBILITY:
Inclusion Criteria

* Female patients must be of non-childbearing potential
* Recent acute coronary syndrome [(ACS) ST elevation myocardial infarction (STEMI), non-STEMI or unstable angina) event documented by ECG, cardiac enzymes or angiogram] 1 - 3 months prior to randomization
* Carotid or ascending aorta artery plaque inflammation Target-to-Background Ratio (TBR) ≥ 1.6
* Receiving concomitant statin therapy following the qualifying ACS event for a minimum of 4 weeks, including a stable statin dose regimen for 2 weeks prior to randomization.

Exclusion Criteria

* Renal insufficiency defined as creatinine >1.5 x upper limit of normal (ULN)
* Cirrhosis, recent hepatitis, alanine aminotransferase (ALT) >1.5 x ULN (i.e., above the normal range) or positive screening test for hepatitis B (hepatitis B surface antigen) or hepatitis C (by ELISA)
* Type I diabetes and uncontrolled Type 2 diabetes defined as hemoglobin A1c (HbA1c) > 9%
* Heart failure defined by New York Heart Association Class III or IV
* Coronary Artery Bypass Surgery (CABG) within 4 months of randomization
* Use of zileuton, montelukast, coumadin or steroids
* Acetaminophen use in any form in the 7 days before enrollment at Visit 1
* Allergy to contrast agents
* Planned additional cardiac intervention (e.g., PCI, CABG) within next 6 months
* Current atrial fibrillation, atrial flutter or frequent premature ventricular contractions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Taub, MD, Study Director — VIA Pharmaceuticals
Locations (2):
- United States (2):
  - VIA Pharmaceuticals, San Francisco, California
  - VIA Pharmaceuticals, Princeton, New Jersey

REFERENCES:
- [Derived] Gaztanaga J, Farkouh M, Rudd JH, Brotz TM, Rosenbaum D, Mani V, Kerwin TC, Taub R, Tardif JC, Tawakol A, Fayad ZA. A phase 2 randomized, double-blind, placebo-controlled study of the effect of VIA-2291, a 5-lipoxygenase inhibitor, on vascular inflammation in patients after an acute coronary syndrome. Atherosclerosis. 2015 May;240(1):53-60. doi: 10.1016/j.atherosclerosis.2015.02.027. Epub 2015 Feb 24. PMID 25752438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened between November 2007 and April 2009
Pre-assignment Details: Subjects had Acute Coronory Syndrome (ACS) 1-3 months prior to randomization and must have received concomitant statin therapy for a minimum of 4 weeks and had a stable statin dose regimen for 2 weeks prior to randomization.
Period: Overall Study
Arm/Group | VIA-2291 | Placebo
Started | 26 | 26
Completed | 24 | 21
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal of consent | 0 | 1
Not completed — Subject returned to home country | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIA-2291 | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 40
  >=65 years | 5 | 7 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 56.2 (9.50) | 58.7 (8.00) | 57.4 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31
  Canada | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plaque Imaging After 24 Weeks
Description: To evaluate the effect of VIA-2291 100 mg relative to placebo on the change from baseline in the target (plaque) to background (blood) ratio (TBR) from an index vessel (either right carotid, left carotid or ascending aorta) based on the standardized 18fluorodeoxy glucose (FDG) uptake measured with PET in patients with acute coronary syndrome and vascular inflammation after 24 weeks of daily dosing.
Time Frame: Baseline and 24 Weeks
Population: Evaluable Population
Measure: Least Squares Mean (95% Confidence Interval); unit: TBR
Arm/Group | VIA-2291 | Placebo
Number analyzed (Participants) | 24 | 21
TBR | -0.01 (11.19) [-0.08 to 0.06] | -0.06 (11.92) [-0.14 to 0.02]
Statistical Analysis 1: Comparison: VIA-2291 vs Placebo; ANCOVA model adjusted for baseline value; Test type: Superiority or Other; p = 0.34, ANCOVA

2. Secondary Outcome: Change From Baseline in Plaque Imaging After 6 Weeks
Description: To evaluate the effect of VIA-2291 100 mg relative to placebo on the change from baseline in the TBR from an index vessel (either right carotid, left carotid or ascending aorta) based on the standardized 18FDG uptake measured with PET in patients after 6 weeks of daily dosing.
Time Frame: Baseline and 6 Weeks
Population: Evaluable Population
Measure: Least Squares Mean (95% Confidence Interval); unit: TBR
Arm/Group | VIA-2291 | Placebo
Number analyzed (Participants) | 24 | 21
TBR | 0.01 (8.37) [-0.07 to 0.08] | -0.07 (9.5) [-0.14 to 0.01]
Statistical Analysis 1: Comparison: VIA-2291 vs Placebo; ANCOVA model adjusted for baseline; Test type: Superiority or Other; p = 0.15, ANCOVA

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | VIA-2291 | Placebo
Serious Adverse Events (participants affected / at risk) | 5/26 | 5/26
Other Adverse Events (participants affected / at risk) | 15/26 | 17/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIA-2291 (N=26) | Placebo (N=26)
Angina Unstable (Cardiac disorders) | 2 | 1
Angina Pectoris (Cardiac disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
In-Stent Coronary Artery Restenosis (Cardiac disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VIA-2291 (N=26) | Placebo (N=26)
Angina Pectoris (Cardiac disorders) | 4 | 3
Sinus Bradycardia (Cardiac disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Chest Pain (General disorders) | 3 | 1
Asthenia (General disorders) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Low Density Lipoprotein Increased (Investigations) | 2 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Influenza (Infections and infestations) | 2 | 1
Hypotension (Vascular disorders) | 2 | 1
Fatigue (General disorders) | 0 | 5
Angina Unstable (Cardiac disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented as a joint, multi-center publication prior to publishing individual site results.